CLINICAL TRIAL: NCT05719818
Title: Dental Care and Initiation of Anti-osteoporotic Therapy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Rhumato04
Record Dates: First submitted 2022-12-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-11

CONDITIONS: Dental Condition; Osteoporosis
MeSH Terms: conditions — Tooth Diseases; Osteoporosis | interventions — Diphosphonates; Dental Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment initiation: patients with a satisfactory oral assessment authorizing the immediate prescription of treatment.
  Interventions: Drug: biphosphonates
- Surgical dental care: patients requiring surgical dental care before treatment initaition.
  Interventions: Procedure: Dental care

INTERVENTIONS:
Drug: biphosphonates — Initiation of bisphosphonate therapy
  Groups: Treatment initiation
Procedure: Dental care — Surgical dental care
  Groups: Surgical dental care

SUMMARY:
The initiation of bisphosphonate therapy for osteoporosis requires an assessment of the oral status to prevent the risk of osteonecrosis of the jaw. This recommendation is sometimes a hindrance to the initiation of treatment or may be responsible for a delay in treatment or even the failure to initiate treatment. However, in the case of a severe osteoporotic fracture (femoral or humeral neck fracture, vertebral fracture or pelvic fracture), treatment must be rapid because of the major risk of refracture in the short term (multiplied by 5 in the 2 years following the fracture).

In the rheumatology department of the Nice University Hospital, the investigator team take care of patients with osteoporotic fractures either directly in hospital or referred by the orthopedics department as part of a care program. For these patients, the team perform an etiological assessment, bone densitometry and evaluation of the oral status with dental panoramic and tele-expertise to determine if there is an indication to perform surgical care before starting the treatment.

Therefore, the investigator aimed to describe the number of patients requiring dental surgery befor the initiation of bisphosphonate or denosumab treatment before to introduce treatment for osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* osteoporotic fracture requiring treatment with bisphosphonate or denosumab

Exclusion Criteria:

* osteoporotic fracture requiring teriparatide treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the rhumatologic department - Nice University hospital for osteoporotic fracture and for who the treatment, either bisphosphonate or denosumab, has justified a dental evaluation
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Number of patients requiring surgical dental care | 15 months
  describe the number of patients requiring surgical dental care before to start osteoporosis treatment vs the number of patients with a satisfactory oral assessment authorizing the immediate prescription of treatment

SECONDARY OUTCOMES:
Impact of dental care on osteoporosis treatment | Change from baseline
  Delay of treatment implementation (in days)
Impact of dental care on osteoporosis treatment | Change from baseline
  New osteoportic fracture occurence (in day since treatment start)
Impact of dental care on osteoporosis treatment | Change from baseline
  Dental complications apperance

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, CHUN, France

IPD SHARING:
Plan to Share IPD: No
Not scheduled